CLINICAL TRIAL: NCT07231159
Title: Building on Trust: Navigating Preventive Lung, Breast, and Prostate Cancer Screenings at Community Resource Spots
Status: Recruiting | Type: Observational
Sponsor: AdventHealth (Other)
Collaborators: Florida Department of Health (Other Government)
Responsible Party: Sponsor
Other Study IDs: 2343026; 333 (Other Grant/Funding Number: Florida Department of Health)
Record Dates: First submitted 2025-11-14; First posted 2025-11-17 (Actual); Last update posted 2025-11-17 (Actual); Status verified 2025-09

CONDITIONS: Breast Cancer; Lung Cancer (Diagnosis); Prostate Cancer
MeSH Terms: conditions — Breast Neoplasms; Lung Neoplasms; Disease; Prostatic Neoplasms | interventions — Referral and Consultation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- community-based initiative for screening, diagnosis, and treatment of breast, lung, and prostate: Identify differences between adults who accept or decline cancer follow-up diagnosis and treatment, and clinical trial screening Identify barriers and facilitators to cancer screening, diagnosis, treatment, and clinical trial screening Understand perceptions towards navigators in the cancer care continuum
  Interventions: Behavioral: referral for definitive diagnosis based on their cancer screening results
- Recruitment of Stakeholder: Investigators will establish relationships with community stakeholders, providers, and other key personnel to inform them of the program, the study, and opportunities to engage in stakeholder focus groups to provide feedback about program operations. For those interested in participating, a study team member will explain the study and the requirements for participation, review the informed consent form in detail, and obtain consent.
  Interventions: Behavioral: Engagement

INTERVENTIONS:
Behavioral: referral for definitive diagnosis based on their cancer screening results — Need for radiological diagnosis
  Groups: community-based initiative for screening, diagnosis, and treatment of breast, lung, and prostate
Behavioral: Engagement — Engage in stakeholder focus groups to provide feedback about program operations
  Groups: Recruitment of Stakeholder

SUMMARY:
To evaluate a community-based outreach initiative for screening, diagnosis, and treatment of breast, lung, and prostate cancers in underserved adults using the Reach, Effectiveness, Adoption, Implementation, Maintenance (RE-AIM) implementation science framework.

ELIGIBILITY:
Inclusion Criteria:

1. Adult aged 18 or older
2. Seeking care at a CRS or emergency department
3. Meets criteria for lung, breast, and/or prostate cancer screening, as outlined below:

   1. Lung cancer: Adults aged 50 to 80 years who have a 20 pack-year smoking history and currently smoke or have quit within the past 15 years
   2. Breast cancer: Women aged 40 to 74 years
   3. Prostate cancer: Men aged 55 to 69 years
4. Receives a positive screening result for lung, breast, and/or prostate cancer at a study site

Exclusion Criteria:

1. Displays behavior disruptive to other patients or staff
2. Refusal to accept screening for breast, lung, and/or prostate cancers

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Community Resource Spots, Emergency Departments and Urgent Care Centers
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2025-11-17 (Estimated); Primary Completion 2026-08-30 (Estimated); Study Completion 2026-08-31 (Estimated)

PRIMARY OUTCOMES:
The categorization of the RE-AIM model dimensions of Reach, Effectiveness, Adoption, Implementation, and Maintenance, | From enrollment to the end of the 3 month follow-up for a total of 12 months
  Reach will assess the percentage and characteristics of patients screened or excluded, as well as participant versus non-participant profiles.
  Effectiveness will measure the proportion of positive screens referred for confirmatory diagnostics and compare screening rates to Healthy People 2030 goals.
  Adoption will track provider education on breast, lung, and prostate cancer screening guidelines, uptake of screening practices, and staff engagement with navigation programs.
  Implementation will evaluate referrals to navigation, screening rates, and for positive screens: referral time, diagnostic barriers, treatment uptake, and clinical trial screening.
  Maintenance will examine primary outcomes at three months, progress toward HP2030 goals, attrition rates, and differences by patient characteristics.

SECONDARY OUTCOMES:
PROMIS Global Health (HR-QoL) scale | From enrollment to the end of the 3 month follow-up for a total of 12 months
  A 10-item scale to assess physical, mental, and social health on a scale of 5 (Excellent) to 1 (Poor), ability to carry out everyday activities on a scale of 5 (Completely) to 1 (Not at all), emotional problems on a scale of 5 (Never) to 1 (Always), fatigue on a scale of 5 (None) to 1 (Very severe), and pain on a scale of 0 (No pain) to 10 (Worst imaginable pain)
Patient Satisfaction with Logistical Aspects of Navigation Scale (PSN-L) | From enrollment to the end of the 3 month follow-up for a total of 12 months
  A 26-item scale to assess satisfaction with the navigation program on a scale of 3 (Very satisfied) to 1 (Not Satisfied)

CONTACTS AND LOCATIONS:
Overall Officials: Mark Socinski, MD, Principal Investigator — AdventHealth
Locations (1):
- Adventhealth, Orlando, Florida, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kumar AJ, Banco D, Steinberger EE, Chen J, Weidner R, Makim S, Parsons SK. Time to diagnostic resolution after an uncertain screening mammogram in an underserved population. Cancer Med. 2020 May;9(9):3252-3258. doi: 10.1002/cam4.2970. Epub 2020 Mar 11. PMID 32160406
- [Background] Holtrop JS, Rabin BA, Glasgow RE. Qualitative approaches to use of the RE-AIM framework: rationale and methods. BMC Health Serv Res. 2018 Mar 13;18(1):177. doi: 10.1186/s12913-018-2938-8. PMID 29534729
- [Background] Hays RD, Bjorner JB, Revicki DA, Spritzer KL, Cella D. Development of physical and mental health summary scores from the patient-reported outcomes measurement information system (PROMIS) global items. Qual Life Res. 2009 Sep;18(7):873-80. doi: 10.1007/s11136-009-9496-9. Epub 2009 Jun 19. PMID 19543809
- [Background] Carle AC, Jean-Pierre P, Winters P, Valverde P, Wells K, Simon M, Raich P, Patierno S, Katz M, Freund KM, Dudley D, Fiscella K. Psychometric evaluation of the patient satisfaction with logistical aspects of navigation (PSN-L) scale using item response theory. Med Care. 2014 Apr;52(4):354-61. doi: 10.1097/MLR.0000000000000089. PMID 24848207
- [Result] Chen M, Wu VS, Falk D, Cheatham C, Cullen J, Hoehn R. Patient Navigation in Cancer Treatment: A Systematic Review. Curr Oncol Rep. 2024 May;26(5):504-537. doi: 10.1007/s11912-024-01514-9. Epub 2024 Apr 6. PMID 38581470
- [Result] Braun, V., Clarke, V. (2006). Using thematic analysis in psychology. Qualitative Research in Psychology, 3, 77-101
- [Result] Bell-Brown A, Watabayashi K, Delaney D, Carlos RC, Langer SL, Unger JM, Vaidya RR, Darke AK, Hershman DL, Ramsey SD, Shankaran V. Assessment of financial screening and navigation capabilities at National Cancer Institute community oncology clinics. JNCI Cancer Spectr. 2023 Aug 31;7(5):pkad055. doi: 10.1093/jncics/pkad055. PMID 37561111

DOCUMENTS (1):
  • Study Protocol (2025-07-17): https://cdn.clinicaltrials.gov/large-docs/59/NCT07231159/Prot_000.pdf